CLINICAL TRIAL: NCT07025746
Title: Acute Effects of Gastrocnemius Myofascial Release on Cervical Flexion and Extension Range of Motion in Healthy Adults: A Randomized Controlled Trial
Brief Title: Acute Effects of Gastrocnemius Myofascial Release on Cervical Flexion and Extension Range of Motion in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Principal Investigator, Ricardo Cardoso, Phd, University Fernando Pessoa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ESS/LFST-706/25-2
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): A myofascial release technique will be performed using a foam roller (Blackroll Standard, 30 x 15 cm) on the dominant lower limb.
  For the Intervention Group (IG), the technique will be applied to the gastrocnemius muscles. In this group, participants will adopt a semi-seated position on a mat, supported by their arms while keeping the body well aligned. The movement will be performed in the direction of the muscle fibers (cephalocaudal), ensuring the accuracy of the technique.
  The foam roller will be in contact with the targeted muscle, and the participant will apply pressure until experiencing slight discomfort. In this way, a self-massage will be performed following the direction of the muscle fibers.
  Interventions: Device: Dynamic foam rolling
- Control group (No Intervention): The participants will remain at rest in a chair for 4 minutes.

INTERVENTIONS:
Device: Dynamic foam rolling — The foam roller will be in contact with the muscle being tested and the patient will exert a load until they feel a slight pain. In this way, the patient performs a self-massage in the direction of the muscle fibers.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to verify the immediate effects of gastrocnemius myofascial release on the active cervical flexion and extension range of motion.

DETAILED DESCRIPTION:
After completing the questionnaire, 91 healthy participants will be randomly divided into two groups: the Intervention Group (IG) (n=46) and the Control Group (CG) (n=45). In the first assessment (M0), the range of motion of cervical flexion and extension will be measured using a smartphone (Galaxy S21 FE 5G, Android) and the Clinometer application. The myofascial release technique (foam roller) will be applied to the gastrocnemius of the dominant lower limb for 4 minutes (3 sets of 1 minute with 30 seconds of rest). Participants in the control group will remain at complete rest for a period of 4 minutes, lying in the supine position, without performing any type of active or passive intervention. Immediately after the intervention/control, all groups will be reassessed (M1).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of both sexes aged 18-40 years.

Exclusion Criteria:

* Deformities in the lower quadrant region of the body;
* Complaints in this region in the last 6 months;
* Surgical procedures or musculoskeletal, cardiac, renal, metabolic, neurological and or oncological pathologies;
* Limb length discrepancy greater than 1.5 cm;
* Pregnant women;
* Ingestion of non-steroidal anti-inflammatory drugs or consumption of any type of narcotic drugs and participants who have drunk alcohol in the last 12 hours.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-07-04 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of active cervical range of motion in flexion and extension. | Change from Baseline (M0) to Immediately after intervention or control (M1)
  Data will be collected at two time points: baseline assessment (M0) and after the intervention/control (M1).
  Participants will be instructed to sit with their spine straight and supported against the backrest of the chair, with ankles, knees, and hips positioned at 90 degrees. Arms will remain crossed over the chest to prevent compensatory thoracic movements.
  Before the test begins, each participant will be asked to actively perform the flexion and extension movements to the limit of their range of motion, aiming to reduce stiffness and promote familiarization with the assessment protocol.
  Measurements will be taken three times for each movement (active flexion and extension), with 30-second rest intervals between each measurement. The average of the three values will be calculated and recorded as the final value.